CLINICAL TRIAL: NCT02701400
Title: A Randomized Study of Tremelimumab Plus Durvalumab Combination With or Without Radiation in Relapsed Small Cell Lung Cancer
Brief Title: Tremelimumab and Durvalumab With or Without Radiation Therapy in Patients With Relapsed Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Principal Investigator, Taofeek K. Owonikoko, Principal Investigator, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00086004; NCI-2016-00026 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); ESR-14-10531 (Other: AstraZeneca); Winship3112-15 (Other: Emory University/Winship Cancer Institute)
Record Dates: First submitted 2016-02-23; First posted 2016-03-08 (Estimated); Results first posted 2021-06-22 (Actual); Last update posted 2021-06-22 (Actual); Status verified 2021-05

CONDITIONS: Recurrent Small Cell Lung Carcinoma
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — durvalumab; Radiation Dose Hypofractionation; Radiosurgery; tremelimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (tremelimumab, durvalumab) (Experimental): Patients receive tremelimumab IV over 1 hour on day 1. Treatment repeats every 4 weeks for up to 4 courses in the absence of disease progression or unacceptable toxicity. Patients also receive durvalumab IV over 1 hour on day 1. Treatment repeats every 4 weeks for up to 1 year in the absence of disease progression or unacceptable toxicity. Patients achieving disease control may restart treatment upon evidence of progressive disease, with or without confirmation.
  Interventions: Biological: Durvalumab; Biological: Tremelimumab
- Arm II (RT, tremelimumab, durvalumab) (Active Comparator): Patients undergo stereotactic body radiation therapy (SBRT) or hypofractionated radiation therapy daily for 5 days over 1 week or for 3 fractions every other day for 1 week and then receive the same treatment as in Arm I.
  Interventions: Biological: Durvalumab; Radiation: Hypofractionated Radiation Therapy; Radiation: Stereotactic Body Radiation Therapy; Biological: Tremelimumab

INTERVENTIONS:
Biological: Durvalumab — Given IV
  Other Names: MEDI4736
Radiation: Hypofractionated Radiation Therapy — Undergo hypofractionated radiation therapy
  Other Names: Hypofractionated Radiotherapy; Hypofractionation
  Arms: Arm II (RT, tremelimumab, durvalumab)
Radiation: Stereotactic Body Radiation Therapy — Undergo SBRT
  Other Names: SBRT
  Arms: Arm II (RT, tremelimumab, durvalumab)
Biological: Tremelimumab — Given IV
  Other Names: Anti-CTLA4 Human Monoclonal Antibody CP-675,206; CP-675,206; Ticilimumab

SUMMARY:
This randomized clinical trial studies how well tremelimumab and durvalumab with or without radiation therapy works in treating patients with small cell lung cancer that has returned after a period of improvement. Monoclonal antibodies, such as tremelimumab and durvalumab, may limit the ability of tumor cells to grow and spread by enhancing immune function. Radiation therapy uses high energy x-rays to kill tumor cells and shrink tumors. Giving tremelimumab and durvalumab together with radiation therapy may lead to improved clinical benefit.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To assess the efficacy (progression free survival [PFS] and objective response rate [ORR]) of combined immune checkpoint inhibitor therapy as treatment for relapsed small-cell lung cancer (SCLC).

SECONDARY OBJECTIVES:

I. To assess the impact of antigen priming using radiation therapy (XRT) on the efficacy of immune checkpoint inhibitors.

II. To determine immune related objective response rate.

III. To estimate overall survival measured as time from randomization to death from any cause.

TERTIARY OBJECTIVES:

I. To characterize tumor infiltrating lymphocytes (TILs) and programmed cell death 1 ligand 1 (PD-L1)/programmed cell death 1 (PD1) expression in paired tumor biopsies at baseline, end of cycle 2 and at the time of progression.

II. To determine dynamic changes in cell free deoxyribonucleic acid (DNA) (cfDNA) and the immunophenotype of peripheral blood repertoire of circulating lymphocytes using multiparameter flow cytometry.

III. To determine changes in circulating cytokine mediators of inflammation and immunity using Luminex assay.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients receive tremelimumab intravenously (IV) over 1 hour on day 1. Treatment repeats every 4 weeks for up to 4 courses in the absence of disease progression or unacceptable toxicity. Patients also receive durvalumab IV over 1 hour on day 1. Treatment repeats every 4 weeks for up to 1 year in the absence of disease progression or unacceptable toxicity. Patients achieving disease control may restart treatment upon evidence of progressive disease, with or without confirmation.

ARM II: Patients undergo radiation therapy daily for 5 days over 1 week or for 3 fractions every other day for 1 week and then receive the same treatment as in Arm I.

After completion of study treatment, patients are followed up periodically.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent and any locally-required authorization (e.g.,) obtained from the subject prior to performing any protocol-related procedures, including screening evaluations
* Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1 or 2
* Hemoglobin ≥ 9.0 g/dL
* Absolute neutrophil count (ANC) ≥ 1.5 x 10⁹/L (≥ 1500 per mm³)
* Platelet count ≥ 100 x 10⁹/L (≥ 100,000 per mm³)
* Serum bilirubin ≤ 1.5 x institutional upper limit of normal (ULN); this will not apply to subjects with confirmed Gilbert's syndrome (persistent or recurrent hyperbilirubinemia that is predominantly unconjugated in the absence of hemolysis or hepatic pathology), who will be allowed only in consultation with their physician
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) ≤ 2.5 x institutional upper limit of normal unless liver metastases are present, in which case it must be ≤ 5 x ULN
* Serum creatinine clearance (CL) > 40 mL/min by the Cockcroft-Gault formula or by 24-hour urine collection for determination of creatinine clearance
* Female subjects must either be of non-reproductive potential (i.e., post-menopausal by history: ≥ 60 years old and no menses for ≥ 1 year without an alternative medical cause; OR history of hysterectomy, OR history of bilateral tubal ligation, OR history of bilateral oophorectomy) or must have a negative serum pregnancy upon study entry
* Subject is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up
* Patients must have baseline evaluations performed prior to the first dose of study drug and must meet all inclusion and exclusion criteria
* Patients must have histologically or cytologically confirmed small cell lung cancer
* Patients must have measurable disease, defined as at least one lesion (excluding the lesion for XRT) that can be accurately measured in at least one dimension (longest diameter to be recorded for non-nodal lesions and short axis for nodal lesions) as > 20 mm with conventional techniques or as > 10 mm with spiral computed tomography (CT) scan
* Patient must have failed or found to be intolerant of standard frontline platinum-based regimens and must not have received > 2 prior lines of therapy (nota bene [NB]: retreatment with a platinum-based doublet for sensitive relapse counts as another line therapy; however substitution of cisplatin with carboplatin or vice versa due to toxicity does not count as a separate regimen)
* Negative serum pregnancy test within 48 hours before starting study treatment in women with childbearing potential
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Involvement in the planning and/or conduct of the study (applies to both AstraZeneca staff and/or staff at the study site)
* Previous enrollment or randomization in the present study
* Treatment with an investigational product during the last 2 weeks
* Any previous treatment with a PD1 or PD-L1 inhibitor, including durvalumab or an anti-cytotoxic T-lymphocyte-associated protein 4 (CTLA4), including tremelimumab
* Receipt of the last dose of anti-cancer therapy (chemotherapy, immunotherapy, endocrine therapy, targeted therapy, biologic therapy, tumor embolization, monoclonal antibodies, other investigational agent) ≤ 14 days prior to the first dose of study drug (≤ 7 days or four half-lives, whichever is longer, prior to the first dose of study drug for subjects who have received prior tyrosine kinase inhibitors [TKIs] [e.g., erlotinib, gefitinib and crizotinib] and within 6 weeks for nitrosourea or mitomycin C)
* Mean QT interval corrected for heart rate (QTc) ≥ 470 ms calculated from 3 electrocardiograms (ECGs) using Fredericia's Correction
* Current or prior use of immunosuppressive medication within 28 days before the first dose of durvalumab or tremelimumab, with the exceptions of intranasal and inhaled corticosteroids or systemic corticosteroids at physiological doses, which are not to exceed 10 mg/day of prednisone, or an equivalent corticosteroid
* Any unresolved toxicity (> Common Terminology Criteria for Adverse Events [CTCAE] grade 2) from previous anti-cancer therapy; subjects with irreversible toxicity that is not reasonably expected to be exacerbated by the investigational product may be included (e.g., hearing loss, peripherally neuropathy)
* Any prior grade ≥ 3 immune-related adverse event (irAE) while receiving any previous immunotherapy agent, or any unresolved irAE > grade 1
* Active or prior documented autoimmune disease within the past 2 years; NOTE: subjects with vitiligo, Grave's disease, or psoriasis not requiring systemic treatment (within the past 2 years) are not excluded
* Active or prior documented inflammatory bowel disease (e.g., Crohn's disease, ulcerative colitis)
* History of primary immunodeficiency
* History of allogeneic organ transplant
* History of hypersensitivity to durvalumab or any excipient
* History of hypersensitivity to the combination or comparator agent
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, active peptic ulcer disease or gastritis, active bleeding diatheses including any subject known to have evidence of acute or chronic hepatitis B, hepatitis C or human immunodeficiency virus (HIV), or psychiatric illness/social situations that would limit compliance with study requirements or compromise the ability of the subject to give written informed consent
* Known history of previous clinical diagnosis of tuberculosis
* History of leptomeningeal carcinomatosis
* Receipt of live attenuated vaccination within 30 days prior to study entry or within 30 days of receiving durvalumab or tremelimumab
* Female subjects who are pregnant, breast-feeding or male or female patients of reproductive potential who are not employing an effective method of birth control
* Any condition that, in the opinion of the investigator, would interfere with evaluation of study treatment or interpretation of patient safety or study results
* Symptomatic or uncontrolled brain metastases requiring concurrent treatment, inclusive of but not limited to surgery, radiation and/or corticosteroids
* Subjects with uncontrolled seizures
* Female patients who are pregnant or breastfeeding or male or female patients of reproductive potential who are not willing to employ effective birth control from screening to 180 days after the last dose of durvalumab + tremelimumab combination therapy or 90 days after the last dose of durvalumab monotherapy, whichever is the longer time period
* Patients receiving any other investigational agents for any reason or non-investigational agents administered for the purpose of controlling cancer growth (use of conventional external beam radiation therapy will be allowed during protocol therapy solely for palliation of localized painful lesions or bone lesions at risk of fracture provided the radiation field does not encompass any selected target lesions required for assessment)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2016-04-14 (Actual); Primary Completion 2020-08-07 (Actual); Study Completion 2020-08-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Taofeek Owonikoko, MD, PhD, Principal Investigator — Emory University
Locations (2):
- United States (2):
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Emory University/Winship Cancer Institute, Atlanta, Georgia

REFERENCES:
- [Derived] Pakkala S, Higgins K, Chen Z, Sica G, Steuer C, Zhang C, Zhang G, Wang S, Hossain MS, Nazha B, Beardslee T, Khuri FR, Curran W, Lonial S, Waller EK, Ramalingam S, Owonikoko TK. Durvalumab and tremelimumab with or without stereotactic body radiation therapy in relapsed small cell lung cancer: a randomized phase II study. J Immunother Cancer. 2020 Dec;8(2):e001302. doi: 10.1136/jitc-2020-001302. PMID 33428583
- See also: Journal Manuscript — https://orcid.org/0000-0002-7724-7728

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm I (Tremelimumab, Durvalumab) | Arm II (RT, Tremelimumab, Durvalumab)
Started | 9 | 9
Completed | 9 | 9
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (Tremelimumab, Durvalumab) | Arm II (RT, Tremelimumab, Durvalumab) | Total
Number analyzed (Participants) | 9 | 9 | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 4 | 4 | 8
  >=65 years | 5 | 5 | 10
Age, Continuous [Mean (Standard Deviation); unit: years] — The measure of dispersion data are not available. All efforts were made to obtain these data from the PI and the study documentation.
  years | 70.5 (NA) — There is no standard deviation for this trial | 66.86 (NA) — There is no standard deviation for this trial | 67.76 (NA) — There is no standard deviation for this trial
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 7
  Male | 6 | 5 | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 9 | 9 | 18
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 3 | 3
  White | 8 | 5 | 13
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 9 | 9 | 18

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS)
Description: Time from initiation of therapy to objective disease progress or death
Time Frame: From initiation of systemic therapy to first documented disease progression, assessed through study completion, up to 2 years
Measure: Median (Standard Deviation); unit: months
Arm/Group | Arm I (Tremelimumab, Durvalumab) | Arm II (RT, Tremelimumab, Durvalumab)
Number analyzed (Participants) | 9 | 9
months | 2.1 (0) | 3.3 (28.6)

2. Primary Outcome: Objective Response Rate
Description: Disease response to therapy measured according to RECIST 1.1 criteria
Time Frame: After every 2 cycles of treatment (1 cycle = 4 weeks), assessed through study completion, up to 2 years
Measure: Median (Standard Deviation); unit: months
Arm/Group | Arm I (Tremelimumab, Durvalumab) | Arm II (RT, Tremelimumab, Durvalumab)
Number analyzed (Participants) | 9 | 9
months | 2.76 (3.9) | 2.76 (3.9)

3. Secondary Outcome: Immune-related Objective Response Rate
Description: Disease response to treatment using immune-related response rate (irRR) criteria
Time Frame: Assessed after every 2 cycles (1 cycle = 4 weeks) on treatment; assessed through study completion, up to 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Tremelimumab, Durvalumab) | Arm II (RT, Tremelimumab, Durvalumab)
Number analyzed (Participants) | 9 | 9
Participants | 9 | 9

4. Secondary Outcome: Overall Survival
Description: Time interval from entering the study until death
Time Frame: From randomization until death from any cause, assessed through study completion, up to 2 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm I (Tremelimumab, Durvalumab) | Arm II (RT, Tremelimumab, Durvalumab)
Number analyzed (Participants) | 9 | 9
months | 2.8 [0.8 to 12.4] | 5.7 [1.6 to 14.5]

5. Other Pre Specified Outcome: Change From Baseline in the Proportion of Lymphocyte Subset (CD8+ICOS+) Between Baseline and On-Treament (End of Cycle 1)
Description: Change in circulating and tumor-infiltrating lymphocytes between baseline and on-treatment samples at the end of Cycle 1. The proportion was calculated as the number of specific lymphocytes subset out of the total number of lymphocytes at baseline compared to the same proportion at the end of cycle 1.
Time Frame: Result presented for assessment at baseline and the end of cycle 1.
Population: All patients with at least 2 paired samples collected at baseline and on-treatment at end of cycle 1
Measure: Mean (95% Confidence Interval); unit: proportion of CD8+ICOS+ Tcells
Units Other Than Participants: lymphocyte subtypes
Groups:
- Pooled Analysis (Arms I and II): Durvalumab: Given IV
  Tremelimumab: Given IV
  Patients in Arm II undergo stereotactic body radiation therapy (SBRT) or hypofractionated radiation therapy daily for 5 days over 1 week or for 3 fractions every other day for 1 week and then receive the same treatment as in Arm I.
Arm/Group | Pooled Analysis (Arms I and II)
Number analyzed (Participants) | 8
Number analyzed (lymphocyte subtypes) | 13
proportion of CD8+ICOS+ Tcells | 1.399 [0.03091 to 2.766]

ADVERSE EVENTS:
Time Frame: Adverse events collected through study completion, up to 2 years.
Arm/Group | Arm I (Tremelimumab, Durvalumab) | Arm II (RT, Tremelimumab, Durvalumab)
All-Cause Mortality (participants affected / at risk) | 9/9 | 8/9
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/9
Other Adverse Events (participants affected / at risk) | 0/9 | 0/9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-05-24): https://cdn.clinicaltrials.gov/large-docs/00/NCT02701400/Prot_SAP_000.pdf